CLINICAL TRIAL: NCT06188403
Title: Comparison of Radiographic Accuracy Between Pre-bent Titanium Plates and 3D Customized Titanium Plates After le Fort 1 Osteotomy in Orthognathic Surgery
Brief Title: Comparison Between Prebent Plates and Custom Plates After le Fort 1 in Orthognathic Surgery
Acronym: customortho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Orthognathic2
Record Dates: First submitted 2023-12-09; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Orthognathic Surgery
Keywords: orthognathic; virtual planning; custom plates
MeSH Terms: interventions — Orthognathic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (group one) will be treated with custom titanium plates and guide to reposition the maxilla (Active Comparator): 7 patients are included in this arm. Le Fort I osteotomy using CAD CAM surgical guide and 3Dcustomized plate are placed to reposition the maxilla according to the virtual surgical planning.
  Interventions: Procedure: Orthognathic surgery (lefort1)
- (group 2) will be treated with prebent titanium plates (Active Comparator): 7 patients are included in this arm. le fort 1 osteotomy using surgical guide and pre-bent stock titanium plates are used after their adaptation on the model of postoperative plan.
  Interventions: Procedure: Orthognathic surgery (lefort1)

INTERVENTIONS:
Procedure: Orthognathic surgery (lefort1) — Lefort 1 osteotomy to reposition the maxilla using two different techniques to achieve more accurate results , one with guide for cutting and placing pre bent stock plates and the other method using custom titanium plates with guide for cutting and placing the plate
  Other Names: Dentofacial surgery

SUMMARY:
patients with dentofacial deformities , who needs lefort 1 osteotomy to correct position of maxilla , are divided into two groups: one group receives custom titanium plates which is patient specific and the other group receives prebent titanium plates done on printed postop plan model before surgery.

ELIGIBILITY:
Inclusion Criteria:

* . Patients with non-syndromic dentofacial deformity requiring Le Fort I with or without bimaxillary osteotomy.

Exclusion Criteria:

1. Patients with acute infection at surgery site.
2. Patient with Systemic disorders contraindicating surgery.
3. Smokers.
4. Alcohol or drug abuse is prohibited.
5. patients who suffered from craniofacial syndrome.
6. patients who had previous orthognathic surgery.
7. patients who had previous maxillary or mandibular trauma

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Radiographic accuracy between postoperative plan and postoperative result. | one month
  Cone Beam Computed tomography (CBCT) is used at 1 month to assess surgical outcome by comparing the clinical results with the virtually planned outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Faculty of dentistry, Alexandria, Egypt